CLINICAL TRIAL: NCT00571402
Title: Family-Focused Psychoeducation for Bipolar Adolescents
Brief Title: Evaluating the Effectiveness of Family-Focused Psychoeducation in Treating Adolescents With Bipolar Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH062555 (NIH); R21MH062555 (NIH); DSIR CT-S
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Disorder
Keywords: Family Treatment; Pharmacotherapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFT (Experimental): Family-focused therapy (FFT) and pharmacotherapy for adolescents, a 21 session family psychoeducational interventio0n administered with best practice medication treatment
  Interventions: Behavioral: Family-focused therapy for adolescents
- Echanced Care (Active Comparator): Enhanced care (EC) and pharmacotherapy for adolescents
  Interventions: Behavioral: Enhanced care

INTERVENTIONS:
Behavioral: Family-focused therapy for adolescents — FFT includes 25 sessions of psychoeducation, communication enhancement training, and problem-solving skills training plus ongoing pharmacological maintenance.
  Other Names: FFT-A
  Arms: FFT
Behavioral: Enhanced care — Enhanced care includes 3 sessions of family psychoeducation plus ongoing pharmacological maintenance.
  Other Names: Treatment as usual (TAU)
  Arms: Echanced Care

SUMMARY:
This study will evaluate the effectiveness of family-focused psychoeducational treatment along with medication in treating adolescents with bipolar I disorder.

DETAILED DESCRIPTION:
Bipolar disorder, also called manic-depressive illness, is a brain disorder that causes dramatic changes in a person's mood and energy. People with bipolar disorder undergo periods of extreme happiness and extreme sadness, known as episodes of mania and depression. Early onset of bipolar disorder poses an especially high health risk to affected individuals. For example, adolescents with bipolar I disorder are at increased risk for hospitalizations, social and academic deterioration, suicide, substance abuse, and nonadherence to medications. Treatment-based research for bipolar adolescents has lagged behind research for adults, particularly in the psychosocial arena. Family-focused treatment (FFT), consisting of psychoeducation about bipolar disorder for the patient and relatives, communication enhancement training, and problem-solving training, has shown promise as an effective psychosocial model. In two previous studies, FFT was found to be a useful addition to bipolar medications in treating adult bipolar I disorder. This study will test the effectiveness of FFT that is centered upon the developmental needs of adolescents with bipolar I disorder.

This study will be divided into three phases. In Phases I and II, adolescent participants and their parents will be enrolled into FFT sessions; the adolescents will also be treated with medications using a clinical management manual. The first two phases will be used to revise and perfect the FFT adolescent (FFT-A) focused manual to be used in the Phase III clinical trial portion of the study.

Participation in Phase III will last about 2 years. All adolescent and parent participants in Phase III will first undergo research interviews. Child-only interviews will last 2 hours and will include questions about mood problems, problems with friends or family members, and substance use history. Parent-only interviews will be conducted in two 1-hour sessions and will include questions about their child's mood and behavioral problems, treatments, and how their child's problems have affected family life. Parent participants will also be asked to assist their child in filling out a questionnaire on mood and behavioral problems and to fill out a questionnaire concerning their own history of problems with mood or anxiety. The last of the initial research interviews will be conducted at the University of Colorado's Psychology Department. Parent and child participants, as well as other relatives, will be asked to talk about problems in family life and ways to solve them. Participants will also be asked to describe pictures from inkblot cards.

Next, participants in Phase III will be divided into 1 of 2 treatment groups: FFT-A plus standard bipolar medication or treatment as usual (TAU) plus standard bipolar medication. There will be a total of 25 FFT sessions over a 2-year period. The sessions will occur weekly for 12 weeks, every other week for the next 12 weeks, every month for 3 more months, and every 3 months for 1 more year. During FFT sessions, parent and adolescent participants will learn about mood disorders and ways to solve family problems. The sessions will be held at the Denver Children's Hospital, the University of Colorado Health Sciences Center's outpatient offices, or the University of Colorado's Psychology Department. Participants receiving TAU will be given an educational workbook on mood disorders and ways to cope with them as a family. TAU participants will attend three 3-hour family counseling sessions to explain the content of the workbook. The sessions will take place at the same locations as the FFT sessions. Child participants in both groups will take their prescribed medications for their bipolar disorder and will continue to see their psychiatrists on a regular basis.

Repeat research interviews will occur every 3 months during the first year of the study and every 6 months during the second year of the study. Questionnaires will be distributed for children and their parents every 6 weeks during the first year of the study and every 3 months during the second year of the study. A questionnaire on the child's functioning in the school setting will also be sent to the child participant's school teacher every 3 months. Outcome assessments will be made at baseline and Months 3, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for bipolar I, bipolar II, or not otherwise specified (NOS) disorder based on independent Kiddie Schedule for Affective Disorders and Schizophrenia and on present and lifetime version interviews with the patient and at least one parent
* Concurrent physician diagnosis of bipolar I, II, or NOS disorder based on a separate set of evaluations of the parent and child
* At least a 1-week episode of manic, mixed, or hypomanic symptoms or a 2-week episode of depressive symptoms within the 3 months prior to study entry
* Currently taking or willing to proceed with regular pharmacotherapy from a study psychiatrist
* At least one biological parent or step-parent with whom the patient lives who is willing to participate in treatment

Exclusion Criteria:

* History of severe, unremitting psychosis lasting more than 3 months
* Evidence of mental retardation (IQ less than 70), organic central nervous system (CNS) disorder, or pervasive developmental disorder
* Substance or alcohol dependence or abuse disorders in the 3 months prior to study entry
* Current life-threatening eating disorder or medical disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2001-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Adolescent Longitudinal Interval Follow-up Examination | Measured at baseline and Months 3, 6, 9, and 12

SECONDARY OUTCOMES:
Kiddie Schedule for Affective Disorders and Schizophrenia | Measured at baseline and Months 3, 6, 9, and 12
Depression and Mania Rating Scales | Measured at baseline and Months 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: David J. Miklowitz, PhD, Principal Investigator — University of Colorado at Boulder; David A. Axelson, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Department of Psychology, University of Colorado, Boulder, Colorado
  - Child and Adolescent Bipolar Services Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Miklowitz DJ, George EL, Axelson DA, Kim EY, Birmaher B, Schneck C, Beresford C, Craighead WE, Brent DA. Family-focused treatment for adolescents with bipolar disorder. J Affect Disord. 2004 Oct;82 Suppl 1(Suppl 1):S113-28. doi: 10.1016/j.jad.2004.05.020. PMID 15571785
- [Background] Miklowitz DJ, Biuckians A, Richards JA. Early-onset bipolar disorder: a family treatment perspective. Dev Psychopathol. 2006 Fall;18(4):1247-65. doi: 10.1017/S0954579406060603. PMID 17064437
- [Result] Miklowitz DJ, Axelson DA, Birmaher B, George EL, Taylor DO, Schneck CD, Beresford CA, Dickinson LM, Craighead WE, Brent DA. Family-focused treatment for adolescents with bipolar disorder: results of a 2-year randomized trial. Arch Gen Psychiatry. 2008 Sep;65(9):1053-61. doi: 10.1001/archpsyc.65.9.1053. PMID 18762591
- [Result] Miklowitz DJ, Axelson DA, George EL, Taylor DO, Schneck CD, Sullivan AE, Dickinson LM, Birmaher B. Expressed emotion moderates the effects of family-focused treatment for bipolar adolescents. J Am Acad Child Adolesc Psychiatry. 2009 Jun;48(6):643-651. doi: 10.1097/CHI.0b013e3181a0ab9d. PMID 19454920